CLINICAL TRIAL: NCT06631885
Title: Efficacy of Integrated Nano-technology in the Irrigation Protocol of Revascularization Technique In Immature Necrotic Teeth (Randomized Clinical Trial)
Brief Title: Efficacy of Integrated Nano-technology in Revascularization of Immature Necrotic Teeth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mohammed abdelmawla mohammed, assisstant lecturer of endodontics, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (586/2022)
Record Dates: First submitted 2024-09-13; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Immature Teeth; Necrotic Pulp
Keywords: regenerative endodontic procedure
MeSH Terms: conditions — Dental Pulp Necrosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group: using AAE protocol (Active Comparator): revascularization using blood clot according to the standardized protocol of the American association of endodontics
  Interventions: Procedure: regenerative endodontic procedure using blood clot according to AAE
- test group (Experimental): diode laser will be used to activate photosensitized nano chitosan 2% for canal disinfection instead of NaOCl in the first visit of revascularization protocol
  Interventions: Procedure: regenerative endodontic procedure using photo activated nanochitosan 2%

INTERVENTIONS:
Procedure: regenerative endodontic procedure using blood clot according to AAE — regenerative endodontic procedure using blood clot to replace the necrotic pulp tissues in immature teeth with a pulp like to tissue to complete root development. using AAE protocol
  Arms: control group: using AAE protocol
Procedure: regenerative endodontic procedure using photo activated nanochitosan 2% — regenerative endodontic procedure using blood clot to replace the necrotic pulp tissues in immature teeth with a pulp like to tissue to complete root development. using photosensitized nanochitosan for root canal disinfection
  Arms: test group

SUMMARY:
This trial aims to study the effect of photoactivated disinfection using Diod laser (810 nm) to activate photosensitive nanoparticle chitosan as an endodontic irrigant versus sodium hypochlorite followed by saline and then EDTA 17% on 1) postoperative pain and 2) the success of revascularization in patients with necrotic immature maxillary anterior teeth using a randomized clinical trial design.

DETAILED DESCRIPTION:
randomized clinical trial will be conducted to investigate and compare the efficacy of photosensitized nano-chitosan 2% as an endodontic disinfectant during revascularization versus sodium hypochlorite, followed by EDTA 17% according to the standardized protocol of the American Association of endodontics.

Twenty individuals with necrotic, immature permanent anterior teeth will be recruited. They will be randomly assigned into two groups according to the received intervention: control group and test group.

pain will be evaluated as a primary outcome at 24 hours and one week post-intervention using numerical rating scale (NRS). In addition, the root development in terms of change in root length and apical foramen diameter and periapical bone healing will be evaluated as secondary outcomes using cone beam tomography.

ELIGIBILITY:
Inclusion Criteria:

* o Immature necrotic maxillary incisor with open apex greater than 1 mm.

  * Teeth where pulp space are not needed for post and core.
  * A restorable tooth.
  * Patients should be free from any systemic disease that may affect normal healing and predictable outcome.
  * Patients who will agree to the consent and will commit to follow-up period.

Exclusion Criteria:

* o Non-restorable teeth.

  * Teeth with root fractures, internal or external root resorption.
  * Teeth with mature fully developed root with closed apex
  * Patients with any systemic disease that may affect predictable outcome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-11 (Estimated); Primary Completion 2024-11-11 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
pain intensity assessed by numerical rating scale | 24 hours and 1 week after completion of the procedure
  postoperative pain using numerical rating scale

SECONDARY OUTCOMES:
root development | 6 months, 1 year postoperative
  change of root length
Apical foramen closure | 6 months, 1 year postoperative
  change in apical foramen diameter
periapical bone healing | 6 months, 1 year postoperative
  change in the area of periapical lesion

IPD SHARING:
Plan to Share IPD: No